CLINICAL TRIAL: NCT01995799
Title: ASSESSMENT OF CELLULAR INFLAMMATION FOLLOWING ACUTE MYOCARDIAL INFARCTION Application Of Ultrasmall Superparamagnetic Particles Of Iron Oxide
Brief Title: IRon Nanoparticle Enhanced MRI in the Assessment of Myocardial infarctioN
Acronym: IRNMAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013/R/CAR/04
Record Dates: First submitted 2013-06-19; First posted 2013-11-27 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Myocardial Infarction; Inflammation
Keywords: Myocardial Infarction (and related inflammation)
MeSH Terms: conditions — Myocardial Infarction; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- USPIO timepoint 2-4 days (Experimental): USPIO given 2-4 days post MI Ferumoxytol enhanced MRI
  Interventions: Device: Ferumoxytol enhanced MRI
- USPIO timepoint 5-7 days (Experimental): USPIO given 5-7 days post MI Ferumoxytol enhanced MRI
  Interventions: Device: Ferumoxytol enhanced MRI
- USPIO tiempoint 11-21 days (Experimental): USPIO given 11-21 days post MI Ferumoxytol enhanced MRI
  Interventions: Device: Ferumoxytol enhanced MRI

INTERVENTIONS:
Device: Ferumoxytol enhanced MRI — Ferumoxytol enhanced MRI scan

SUMMARY:
Ferumoxytol is an example of a 'smart' magnetic resonance contrast agent that consists of ultrasmall superparamagnetic particles of iron oxide (USPIOs) and is avidly taken up by macrophages. Through a previous work, the investigators have established that USPIOs can identify inflammation in the wall of abdominal aortic aneurysms and that this is associated with a three-fold increase in the rate of aneurysm growth. The utility of ferumoxytol for imaging cardiovascular inflammation in other areas of the body has yet to be established but Dr Alam has established uptake of USPIOs in the penumbra and infarct zone of the myocardium in patients with a recent myocardial infarction. The investigators wish to assess USPIO uptake in patients with recent acute myocardial infarction and identify the time course and determinants of cellular tissue inflammation. This will be the first clinical study to examine the ability of USPIOs to image myocardial inflammation following acute myocardial infarction.

DETAILED DESCRIPTION:
Background

Coronary atherosclerosis is responsible for the initiation of acute myocardial infarction with plaque rupture leading to acute coronary thrombosis and myocardial infarction. Current treatment in the acute phase involves re-establishing vessel patency by percutaneous coronary intervention supported by anti-thrombotic therapy. Thereafter, statins, angiotensin-converting enzyme inhibitors and beta-blockade all have prognostic benefit but no treatments have been successfully developed to target post-infarction inflammatory pathways.

Necrotic cardiac muscle elicits an inflammatory cascade that serves to clear the infarct of dead cells and matrix debris. Human cardiac muscle has negligible regenerative capacity and ultimately inflammation leads to replacement of damaged tissue with a fibrotic scar. Enhancing reparative mechanisms following the inflammatory reaction to myocardial infarction may reduce cardiomyocyte injury, attenuate adverse remodelling and improve clinical outcome. A better understanding of the early post-infarct healing phase will also facilitate cell therapy strategies to engraft stem cells or stimulate regeneration. In order to achieve this goal, the investigators must better characterise the inflammatory processes that follow infarction and myocardial necrosis in humans.

Inflammatory cell mediated injury and healing in the infarcted myocardium

Neutrophils Inflammation within the infarcted myocardium is associated with induction of endothelial adhesion molecules and enhanced permeability of the microvasculature. Up regulation of chemokines including interleukin (IL)-8 and monocyte chemoattractant protein (MCP)-1 attracts neutrophils and monocytes to the site of injury. Early reperfusion therapy amplifies this inflammatory cell influx and accelerates the healing response through proliferative and maturation phases. Neutrophil adhesion to endothelium of infarcted myocardium occurs within minutes of reperfusion. Ischaemic cardiomyocytes are further injured by adherent neutrophils that release reactive oxygen species and destructive proteases including human neutrophil elastase (HNE) and proteinase 3. HNE has a wide range of substrates including matrix components elastin, fibronectin, and collagen types III and IV. Activated neutrophils also occlude microvessels and increase endothelial permeability contributing to myocardial oedema. Capillary plugging and obstruction by activated neutrophils contributes to failure of microvascular perfusion and increased infarct size within the 'no-reflow' zone. Neutrophil depletion reduces this phenomenon and infarct size following reperfusion in pre-clinical models.

Monocyte-derived Macrophages

Recruitment of monocytes into the infarcted myocardium is followed by maturation and differentiation into macrophages: a process dependent on growth factors such as macrophage-colony stimulating factor (M-CSF). Macrophages have multiple roles within the infarct including (i) phagocytic clearance of dead cells and debris, (ii) production of growth factors and cytokines that stimulate fibroblast growth and angioneogenesis, and (iii) matrix turnover through the production of matrix metalloproteases and their inhibitors. Macrophages are resident within 24 h of infarction and persist for up to 4 weeks. During this period, macrophages regulate infarct healing with the initial development of granulation tissue and subsequent scar formation. Murine studies suggest that distinct monocyte subsets regulate these different processes. Monocytes arriving within the first 3 days mature into macrophages that scavenge necrotic debris through inflammatory mediator expression, proteolysis and phagocytosis while monocytes arriving later on give rise to macrophages which promote reparative processes such as angioneogenesis and extracellular matrix deposition. Apoptosis is the primary mechanism determining longevity of neutrophils within sites of inflammation and infarction. Engulfment and clearance of apoptotic neutrophils by macrophages produces potent anti-inflammatory signals including release of transforming growth factor (TGF)-β. Combined with clearance of pro-inflammatory matrix fragments, these processes drive the switch to tissue repair and resolution of the post-infarct inflammatory response.

MCP-1 expression is increased in ischaemic myocardium following reperfusion and this accounts for a substantial proportion of the monocyte chemotactic activity. MCP-1 knockout mice exhibit delayed macrophage infiltration in the healing infarct with a prolonged inflammatory phase and delayed replacement of injured cardiomyocytes with granulation tissue. The MCP-1 deficient mice have similar size infarcts but attenuated remodelling compared to wild types. MCP-1 mRNA levels are increased 40-fold within non-infarcted myocardium and blockade of MCP-1 signalling with a deletion mutant of MCP-1 markedly reduced macrophage infiltration both within the infarct and non-infarcted myocardium. Widespread myocardial inflammatory cell infiltration beyond the non-infarcted zone has been observed in human autopsy specimens. Blockade of MCP-1 signalling is associated with improved survival rates and reduced left ventricular dilatation as well as reduced tumour necrosis factor (TNF)-α gene expression in the non-infarcted myocardium. These studies indicate that macrophage activity outside the infarct zone may contribute to adverse myocardial remodelling following myocardial infarction.

The inflammatory response to myocardial infarction is necessarily complex to coordinate the development of a healing scar from infarcted tissue. The role of the macrophage differs depending on differentiation and location within the myocardium. Therapeutic manipulation of this healing process will only come from understanding mechanisms and targeting reparative pathways. Indiscriminate immunosuppressive therapy in this setting may result in harm as observed in trials with methylprednisolone in acute myocardial infarction.

Magnetic Resonance Imaging in Tracking Cellular Inflammation

Iron oxide particles can be used as a contrast medium in magnetic resonance imaging since they can alter the magnetic properties and relaxation of tissues after application of radiofrequency pulses. Such contrast media consist of an iron oxide core within a dextran coat. They can be classified as "superparamagnetic iron oxide particles" (SPIOs) consisting of particles over 30 nm in diameter, or "ultrasmall superparamagnetic iron oxide particles" (USPIOs) which are under 30 nm in diameter. USPIOs are taken up by cells of the liver, spleen, bone marrow and lymph nodes. They have the capacity to extravasate through capillaries and be phagocytosed by tissue inflammatory cells of the reticuloendothelial system. These cells are predominately macrophages, but neutrophils have also been shown to take up USPIOs. This model of USPIO-enhanced MRI can highlight areas of inflammation in models of vertebral osteomyelitis, aortic atherosclerosis, arthritis-induced hyperperfusion, autoimmune encephalomyelitis, nephritis and nephropathy, cerebral ischaemia and renal ischaemia.

Pilot Data in Patients With Acute Myocardial Infarction

The investigators have undertaken preliminary proof-of-concept studies examining the possibility of using USPIOs to image the myocardium in patients having sustained a recent acute myocardial infarction. To date, the investigators have studied 16 patients following ST segment elevation myocardial infarction treated with reperfusion therapy and undertaken serial magnetic resonance imaging scans. By undertaking T2* maps of the myocardium before and 24-h after USPIO administration, the investigators calculated the R2* value (the inverse of T2*) and represented this as a colour-coded R2* map. This demonstrated a 2-3 fold increase in the R2* value in the infarct and peri-infarct area. As a negative control, the investigators have observed little or no change in the R2* value in myocardium remote from the site of ischaemia or skeletal muscle. The liver demonstrates marked uptake of USPIOs with a 3-4 fold increase in R2* value.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Plasma troponin concentration >5 ng/mL; upper limit of normal 0.04 ng/mL)
* Acute myocardial infarction defined according to the Universal Definition of myocardial infarction

Exclusion Criteria:

* Critical (≥95%) left main stem coronary artery stenosis
* Continued symptoms of angina at rest or minimal exertion
* Past history of systemic iron overload or haemochromatosis
* Renal failure (estimated glomerular filtration rate <25 mL/min)
* Contraindication to magnetic resonance imaging
* Significant heart failure (Killip class ≥2)
* Known allergy to dextran- or iron-containing compounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05-24 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
R2* value | MRI 24 hrs after USPIO infusion (regardless of time-point given)
  Marker of USPIO uptake (and inflammation) in each cohort after myocardial infarction.
  The USPIO infusion is given at different time-points for each cohort. However only the R2* value on the MRI 24 hours after infusion will constitute the primary end-point

SECONDARY OUTCOMES:
Serum Inflammatory markers | 2-104 days post MI
  Correlation between blood and MRI inflammatory markers

OTHER OUTCOMES:
MRI parameters | 2-104 days
  Ejection fraction change over time
MRI parameters | Baseline and 3 months
  Late enhancement volume change
MRI parameter | Baseline
  T2 oedema

CONTACTS AND LOCATIONS:
Overall Officials: Shirjel R Alam, MBChB, Study Director — University of Edinburgh
Locations (2):
- United Kingdom (2):
  - Royal Infirmary of Edinburgh, Edinburgh, Lothian
  - Clinical Research Imaging Centre, Edinburgh, Lothian